CLINICAL TRIAL: NCT00746317
Title: A Phase I, Open-Label, Multi-center, Dose-escalation Study of the Safety, Tolerability, and Pharmacokinetics of GC33 Administered Weekly in Patients With Advanced or Metastatic Hepatocellular Carcinoma (HCC)
Brief Title: A Phase I Study of GC33 in Advanced or Metastatic Liver Cancer (Hepatocellular Carcinoma)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chugai Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GC-001US
Record Dates: First submitted 2008-09-01; First posted 2008-09-03 (Estimated); Last update posted 2012-10-17 (Estimated); Status verified 2012-10

CONDITIONS: Advanced or Metastatic HCC
MeSH Terms: interventions — codrituzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: GC33

INTERVENTIONS:
Drug: GC33 — IV administration at 4 escalating dose levels.

SUMMARY:
This phase I trial is studying the safety and best dose of GC33 in patients with advanced or metastatic liver cancer.

DETAILED DESCRIPTION:
This is a Phase I open-label dose escalation study of GC33 in patients with advanced or metastatic HCC. This study is designed to evaluate safety, tolerability, pharmacokinetics, and preliminary assessment of anti-tumor activity. Enrollment will proceed until a maximum tolerated dose (MTD) and a recommended Phase II dose has been established.

ELIGIBILITY:
Inclusion Criteria:

* Signed written Institutional Review Board (IRB)/Ethical Committee (EC) approved informed consent form
* Male or female ≥ 18 years old.
* Life expectancy ≥ 3 months.
* ECOG Performance Status of 0-1.
* Histologically confirmed hepatocellular carcinoma (without fibrolamellar subtype).
* Not a candidate for curative treatments.
* Child-Pugh A or B.
* Hematological, Biochemical and Organ Function:

  * AST (SGOT): ≤ 5.0 × ULN
  * ALT (SGPT): ≤ 5.0 × ULN
  * Total Bilirubin: ≤ 3.0 × ULN
  * Platelets: ≥ 50,000/μL
  * Absolute Neutrophil Count: ≥ 1,500/μL
  * Serum creatinine: ≤ 2.0 × ULN
  * PT-INR: ≤ 2.0,
* Ability to provide a tumor tissue sample either by:

  * a sample obtained within 3 months prior to informed consent for HCC diagnosis. Resection samples are not acceptable.
  * undergo a biopsy to confirm HCC diagnosis
* At least one measurable lesion based on Response Evaluation Criteria In Solid Tumors criteria.

(Extension Phase)

* Signed written Institutional Review Board (IRB)/Ethical Committee (EC) approved informed consent form.
* Male or female ≥ 18 years old.
* Life expectancy ≥ 3 months.
* ECOG Performance Status of 0-1.
* Histologically confirmed hepatocellular carcinoma (without fibrolamellar subtype).
* Not a candidate for curative treatments.
* Child-Pugh A.
* Hematological, Biochemical and Organ Function:

  * AST (SGOT): ≤ 5.0 × ULN
  * ALT (SGPT): ≤ 5.0 × ULN
  * Total Bilirubin: ≤ 3.0 × ULN
  * Platelets: ≥ 50,000/μL
  * Absolute Neutrophil Count: ≥ 1,500/μL
  * Serum creatinine: ≤ 2.0 × ULN
  * PT-INR: ≤ 2.0
* IHC confirmed GPC3-positive HCC tumor tissue. Tumor tissue sample may be provided by:

  * A formalin fixed paraffin embedded block sample within 12 months prior to informed consent for HCC diagnosis;
  * Unstained slides obtained within 3 months prior to informed consent for HCC diagnosis;
  * Undergo biopsy to confirm GPC3-positive HCC.
  * Resection samples are not acceptable.
* At least one measurable lesion based on Response Evaluation Criteria In Solid Tumors criteria.

Exclusion Criteria:

* Child-Pugh C.
* Pregnant or lactating women or women of child-bearing potential and men of childbearing potential not willing to use effective means of contraception.
* Patients known to be positive for Human immunodeficiency virus infection.
* Active infectious diseases requiring treatment except for hepatitis B and C.
* Other malignancies within the last 5 years.
* History of transplantation (organ, bone marrow transplantation,peripheral blood stem cell transplantation, etc.).
* Patients with significant concomitant disease determined by the investigator to be potentially aggravated by the investigational drug.
* Patients with brain metastases, other central nervous system or other psychiatric disease.
* Patients who received major surgery, local therapy for HCC, chemotherapy, radiotherapy, hormone-therapy, immunotherapy, or another investigational drug within 4 weeks prior to Day 1.
* Patients who received the following treatments within 2 weeks prior to Day1:

  * Anticoagulant or thrombolytic agents for therapeutic purposes.
  * Systemic anti-viral therapy for hepatitis C/cirrhosis.
  * Blood transfusion
* History of hypersensitivity to similar agents.
* Patient is unable to comply with the requirements of the protocol and/or follow-up procedures.

(Extension Phase)

* Child-Pugh B or C.
* Pregnant or lactating women or women of child-bearing potential and men of childbearing potential not willing to use effective means of contraception.
* Patients known to be positive for Human immunodeficiency virus infection.
* Active infectious diseases requiring treatment except for hepatitis B and C.
* Other malignancies within the last 5 years.
* History of transplantation (organ, bone marrow transplantation, Peripheral blood stem cell transplantation, etc.).
* Patients with significant concomitant disease determined by the investigator to be potentially aggravated by the investigational drug.
* Patients with brain metastases, other central nervous system or other psychiatric disease.
* Patients who received major surgery, local therapy for HCC, chemotherapy, radiotherapy, hormone-therapy, immunotherapy, or another investigational drug within 4 weeks prior to Day 1.
* Patients who received the following treatments within 2 weeks prior to Day 1:

  * Anticoagulations or thrombolytic agents for therapeutic purposes.
  * Systemic anti-viral therapy for hepatitis C/cirrhosis.
  * Blood transfusion
* History of hypersensitivity to similar agents.
* Patient is unable to comply with the requirements of the protocol and/or follow-up procedures.
* IHC confirmed GPC3-negative HCC tumor tissue.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2008-09; Primary Completion 2010-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Determine the safety and tolerability of escalating doses of GC33 | Continuously

SECONDARY OUTCOMES:
Characterize the pharmacokinetics of GC33 | Continuously
Perform a preliminary assessment of anti-tumor activity of GC33 | Continuously

CONTACTS AND LOCATIONS:
Overall Officials: Toshihiko Ohtomo, Study Chair — Chugai Pharmaceutical
Locations (9):
- United States (9):
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Center at the Detroit Medical Center, Detroit, Michigan
  - Washington University, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - Methodist Hospital, Houston, Texas
  - Swedish Cancer Institute at the Swedish Medical Center, Seattle, Washington